CLINICAL TRIAL: NCT07181720
Title: Clinical Study of CD70-Targeted Chimeric Antigen Receptor T Lymphocytes (CAR-T) in Advanced CD70-Positive Malignant Solid Tumors
Brief Title: CD70-Targeted CAR-T Therapy in CD70-Positive Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC095
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Renal Cell Carcinoma (RCC); Lung Cancer; Anaplastic Thyroid Carcinomas; Ovarian Cancer; Cervical Cancer; Thymic Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Lung Neoplasms; Thyroid Carcinoma, Anaplastic; Ovarian Neoplasms; Uterine Cervical Neoplasms; Thymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous of CD70-targeted CAR-T (Experimental): Infusion of CD70-targeted CAR-T cells by dose of 3-10x10^5 cells/kg
  Interventions: Biological: CD70-targeted CAR-T cells
- Intrapleural infusion of CD70-targeted CAR-T (Experimental): Infusion of CD70-targeted CAR-T cells by dose of 3-10x10^5 cells/kg
  Interventions: Biological: CD70-targeted CAR-T cells
- Intraperitoneal infusion of CD70-targeted CAR-T (Experimental): Infusion of CD70-targeted CAR-T cells by dose of 3-10x10^5 cells/kg
  Interventions: Biological: CD70-targeted CAR-T cells

INTERVENTIONS:
Biological: CD70-targeted CAR-T cells — Administration method: intravenous infusion. Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.
  Arms: Intravenous of CD70-targeted CAR-T
Biological: CD70-targeted CAR-T cells — Administration method: intrapleural infusion. Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.
  Arms: Intrapleural infusion of CD70-targeted CAR-T
Biological: CD70-targeted CAR-T cells — Administration method: intraperitoneal infusion. Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.
  Arms: Intraperitoneal infusion of CD70-targeted CAR-T

SUMMARY:
This study is a single-arm, open-label, dose-escalating + dose-expansion clinical study, aiming to evaluate the safety and efficacy of CD70-targeted CAR-T cell preparations, and to preliminarily observe the study drug in CD70-positive advanced malignant tumors. The pharmacokinetic characteristics of CAR-T cell preparations for the treatment of patients with CD70-positive advanced malignancies were obtained and the recommended dose and infusion schedule.

DETAILED DESCRIPTION:
According to the different infusion methods, patients will be assigned to three parallel subgroups: intravenous infusion, intrapleural infusion, and intraperitoneal infusion.

Within each subgroup, the study is conducted in two sequential parts:

1. .Part A (dose-escalation): escalation begins at the lowest dose level; 3-6 subjects are enrolled at each dose level;
2. .Part B (dose-expansion): additional subjects are treated at the recommended dose identified in Part A to further evaluate safety and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender;
2. Histologically or cytologically confirmed advanced/metastatic solid tumors (tumors with positive CD70 expression, confirmed histopathological ly with IHC 3+ score);
3. Failed or intolerant to standard second-line treatments (at least one of the following: tyrosine kinase inhibitors (TKIs), poly(ADP-ribose) polymerase inhibitors (PARPi), anti-angiogenic therapy; disease progression or inability to tolerate surgery, chemotherapy, radiotherapy, or targeted therapy);
4. At least one measurable lesion per RECIST 1.1 criteria, with measurable lesions defined as:

   1. Extranodal lesions with a long axis ≥10mm on CT scan;
   2. Lymph node lesions with a short axis ≥15mm on CT scan;
   3. CT slice thickness ≤5mm.
5. ECOG performance status of 0-2 ;
6. Expected survival ≥12 weeks;
7. No history of severe psychiatric disorders;
8. Adequate organ function as defined by the following:

   1. Hematology: White blood cell count >2.0×10⁹/L, neutrophils >0.8×10⁹/L, lymphocytes >0.5×10⁹/L, platelets >50×10⁹/L, hemoglobin >90g/L;
   2. Cardiac: Echocardiogram showing left ventricular ejection fraction (LVEF) ≥50%, and ECG with no significant abnormalities;
   3. Renal: Serum creatinine ≤2.0×ULN;
   4. Hepatic: ALT and AST ≤3.0×ULN (may be relaxed to ≤5.0×ULN in cases with liver tumor infiltration); total bilirubin ≤2.0×ULN (may be relaxed to ≤3.0×ULN in cases with Gilbert's syndrome or liver tumor infiltration);
   5. Oxygen saturation ≥92% without supplemental oxygen;
9. Ability to undergo single or venous blood collection, with no contraindications to cellular collection;
10. Female subjects must agree to use reliable contraception (excluding fertility awareness methods) from the time of informed consent until 1 year after CAR-T cell infusion;
11. Subject or authorized guardian agrees to participate in the trial and signs the informed consent form (ICF), indicating understanding of the trial's purpose and procedures and willingness to participate.

Exclusion Criteria:

1. Prior treatment with anti-CD70 therapies;
2. Active/symptomatic central nervous system (CNS) metastasis or meningeal metastasis: Subjects with treated brain metastases are eligible if treatment was completed ≥4 weeks prior to screening and there is no evidence of progression on imaging;
3. Prior treatments within specified time frames:

   1. Participation in other interventional clinical trials within 3 months before cell infusion (for unapproved drugs, the last dose must be ≥3 months prior; for approved drugs, ≥5 half-lives prior to cell infusion);
   2. Received chemotherapy or targeted therapy within 2 weeks prior to blood collection or within 5 half-lives of the drug (whichever is shorter);
   3. Received >10mg/day prednisone (or equivalent) within 2 weeks prior to blood collection, unless for adrenal replacement or inhaled/local steroids (except for active autoimmune disease);
   4. Received live attenuated vaccines within 4 weeks prior to screening;
4. Active infection requiring systemic treatment or uncontrolled infection within 1 week before screening;
5. History of any other malignancy within the past 3 years, except for treated and stable non-melanoma skin cancer or malignancies treated with curative intent and no evidence of active disease for ≥3 years;
6. Cardiovascular conditions:

   1. NYHA Class III or IV heart failure;
   2. Myocardial infarction or coronary artery bypass graft (CABG) within 6 months prior to screening;
   3. Clinically significant ventricular arrhythmias or unexplained syncope (excluding vasovagal or dehydration);
   4. Severe non-ischemic cardiomyopathy;
7. Active or uncontrolled autoimmune diseases such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, systemic vasculitis, etc.;
8. Positive for HBsAg or HBcAb with elevated HBV DNA in peripheral blood; positive for HCV antibodies with detectable HCV RNA levels; positive for HIV antibodies; positive syphilis test;
9. Toxicity from prior anti-tumor treatments has not resolved to baseline or ≤grade 1, except for alopecia or peripheral neuropathy;
10. History of venous thromboembolism (e.g., pulmonary embolism) requiring ongoing anticoagulation treatment, or meeting one of the following criteria:

    1. Severe bleeding (grade 3 or 4) lasting for ≥30 days;
    2. Post-thrombotic sequelae (e.g., persistent dyspnea and hypoxia) due to venous thromboembolism;
11. Pregnant or breastfeeding women;
12. Other conditions that, in the opinion of the investigator, make the subject unsuitable for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CAR-T cell preparations in the treatment of CD70-positive advanced malignancies [Safety and Tolerability] | 1 month
  Incidence of adverse events during the study, evaluated per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) criteria
Obtained the recommended dose and infusion regimen of CAR-T cells for the treatment of patients with CD70-positive advanced malignancies [Safety and Tolerability] | 1 month
  Dose-limiting toxicity after CD70 CAR-T cell infusion

SECONDARY OUTCOMES:
Assessing disease control rates of CAR-T cell preparations in CD70-positive advanced malignancies [Effectiveness] | 1 and 3 months
  Disease control rate: The proportion of subjects who achieved CR, PR, SD after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
To characterize the in-vivo cellular kinetics of CAR-T cells【pharmacokinetics】 | From infusion through Month 3
  Cmax: maximum observed level of circulating CAR-T cells in peripheral blood after infusion
To characterize the in-vivo cellular kinetics of CAR-T cells【pharmacokinetics】 | From infusion through Month 3
  To determine the time to maximum observed level of circulating CAR-T cells (Tmax)；To estimate AUC0-28d and AUC0-90d for circulating CAR-T cells
To assess the inflammatory response following CAR-T cell infusion | From infusion through Month 3
  Serum levels of inflammation-related markers and cytokines, including but not limited to C-reactive protein (CRP), interleukin-6 (IL-6), and ferritin

OTHER OUTCOMES:
Objective response rate (ORR) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies [Effectiveness] | 2 years
  Objective response rate includes：The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Duration of Response (DOR) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies [Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies [Effectiveness] | 2 years
  PFS will be assessed from the first CD70 CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
Overall survival(OS)of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies [Effectiveness] | 2 years
  OS will be assessed from the first CD70 CAR-T cell infusion to death from any cause (Assessed by investigators based on IRECIST criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Donglai Lv, MD, Principal Investigator — The 901 Hospital of Joint Logistics Support Force of People Liberation Army
Locations (1):
- The 901 Hospital of Joint Logistics Support Force of People Liberation Army, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No